CLINICAL TRIAL: NCT04072224
Title: Evaluation of the Reproducibility of Ablation Volumes at One Month After Microwave Treatment Compared to the Manufacturer's Abacus: on the Kidney, Liver and Lung
Acronym: Ablation
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018/02
Record Dates: First submitted 2019-07-01; First posted 2019-08-28 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hepatic Tumor; Renal Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Microwave thermal ablation (MO) is recognized as an alternative to surgery for the local-regional treatment of primary and secondary hepatic and renal tumors and for secondary pulmonary tumors in patients at anesthetic and/or surgical risk.

Microwaves have a reputation for not producing reproducible ablation volumes with elliptical deformations and risks of over or under processing.

The Covidien manufacturer offers a microwave system that guarantees more spherical and reproducible ablations: Emprint TM ablation system with Thermosphere TM technology (thermal control, field control, wavelength control).

The investigators have 2 years of experience and therefore propose to carry out a first retrospective study, on a cohort of about fifty patients, whose objective will be to compare the volume of in vivo ablation one month after thermo-ablative treatment by microwave of a hepatic, renal or pulmonary tumour with the reference volume announced by the Covidien abacus manufacturer.

Microwave ablation, which is much less studied, is less used because of the low reproducibility of necrosis volumes.

The Covidien manufacturer offers a system that allows ablation volumes that are supposed to be reproducible, which attracted the Nîmes University Hospital during the call for tenders.

To the investigator's knowledge, there are no studies that have evaluated the actual volume of ablation by this system.

DETAILED DESCRIPTION:
The investigators have 2 years of experience and therefore propose to carry out a first retrospective study, on a cohort of about fifty patients, whose objective will be to compare the volume of in vivo ablation one month after thermo-ablative treatment by microwave of a hepatic, renal or pulmonary tumour with the reference volume announced by the Covidien abacus manufacturer.

Microwave ablation, which is much less studied, is less used because of the low reproducibility of necrosis volumes.

The Covidien manufacturer offers a system that allows ablation volumes that are supposed to be reproducible, which attracted the Nîmes University Hospital during the call for tenders.

To the investigator's knowledge, there are no studies that have evaluated the actual volume of ablation by this system.

This is a retrospective monocentric study that divides patients into three groups according to the organ concerned (liver, kidney, lung). It concerns patients with hepatic, renal or pulmonary tumours whose indication for treatment by thermo-ablation has been validated in RCP at the University Hospital of Nîmes.

Each patient was informed of the therapeutic management and was seen in interventional radiology consultation before the expected date of thermo-ablation.

A letter of no objection was sent to each patient prior to treatment. A CT or MRI control imaging is performed one month before the operation, systematically at the University Hospital of Nîmes after a thermo-ablative procedure.

The size of the ablation volume obtained is measured (major axis and minor axis) on this control imaging. This volume will be compared to the ablation volume planned by the manufacturer, depending on the power and duration of the impact chosen according to the size of the tumor (evaluated on the imaging prior to the procedure).

Data stored in Redcap. 50-60 patients included.

ELIGIBILITY:
Inclusion Criteria:

* thermo-ablative treated patients with MO with the Covidian manufacturer
* primary hepatic or renal or secondary hepatic, renal or pulmonary tumor at the University Hospital of Nîmes between June 2016 and June 2018
* diagnosis and size of the tumour established on the basis of tomodensitometric (CT) or magnetic resonance (MRI) imaging.

Exclusion Criteria

* patients with coagulation disorders
* patients with progressive infectious process contraindicating the procedure and/or for whom thermo-ablation equipment other than Covidien has been used

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major patients who have received thermoablative treatment with MO with the Covidian manufacturer of a primary hepatic or renal tumor or secondary hepatic, renal or pulmonary tumor
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Description of volume of in vivo ablation | at one month
  microwave ablation Versus ablation by the Covidien abacus manufacturer

SECONDARY OUTCOMES:
spleen response | at one month
  - Complications rate measured by microwave
liver response | at one month
  Complications rate measured by microwave

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France